CLINICAL TRIAL: NCT07210034
Title: Prognostic Value of HALP Score, Monocytopenia, Hypofibrinogenemia, and AST/ALT Ratio in Patients With Myelodysplastic Syndromes at Assiut University Hospital.
Brief Title: What is the Prognostic Value of HALP Score, Monocytopenia, Hypofibrinogenemia, and AST/ALT Ratio in Patients With Myelodysplastic Syndromes
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Amira Merzek, Resident at internal medicine department, Assiut University
Other Study IDs: HALP-MDS
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Myelo Dysplastic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
to investigate prognostic significance of many factors in MDS including HALP score ( haemoglobin level, albumin level, lymphocyte, platelets), monocytopenia, hyperfibrinogenemia and AST/ALT ratio in patients with MDS at Assiut University Hospital.

And to study overall survival and leukemia free survival rates in MDS patients.

DETAILED DESCRIPTION:
Frequently seen in advanced age, myelodysplastic syndromes (MDS) are a heterogeneous clonal stem cell disorders characterized by ineffective hematopoiesis and having a risk of progression to acute myeloid leukemia (AML). The clinical course of MDS varies considerably, and most patients cannot tolerate intensive treatment approaches due to their advanced age. Accurate diagnosis and reliable prognostic assessment are of critical importance for making individualized clinical decisions in patients with MDS(2). Therefore, prognostic parameters and/or prognostic scoring systems have been developed to distinguish between patient groups differing in median survival time. An ideal prognostic scoring system should contain merely independent prognostic parameters, and the limits of these parameters should be validated, easily identifiable at diagnosis, and cost-effective. The international prognostic scoring system (IPSS), the revised IPSS (IPSS-R), and the World Health Organization (WHO) prognostic scoring system [WPSS] are the most commonly utilized prognostic models (3,4). However, it is considered that many factors, except for the variables in these systems, may also affect the prognosis of MDS5. Immune response and Inflammatory cells have been defined as very important parameters in cancer survival rate(6). In several recent studies, peripheral blood cells, including absolute lymphocyte count (ALC), monocytes, and platelets (Plt), have been reported to be related to higher mortality rates in lymphoma patients(7,8 ) . In recent years, many combinations of infammatory parameters, such as neutrophil-lymphocyte ratio, platelet-lymphocyte ratio, and lymphocyte-monocyte ratio have been used to predict the prognosis in patients with oncological and hematological malignancies (9-11). Nutritional status has also been emphasized in various studies as an important factor affecting the prognosis(11-13). Previous studies have defined a new infammatory index called the hemoglobin, albumin, lymphocyte, and platelet (HALP) score, which is effective in the prognosis of those with kidney, bladder, stomach, small-cell lung, and prostate cancers(14-17). The HALP score is calculated using four laboratory markers (hemoglobin, albumin, lymphocyte, and platelet), which are the biomarkers of nutrition and Inflammation status. In the field of hematology, the prognostic efficiency of the HALP score has been evaluated in a limited number of studies, including in diffuse large B-cell lymphoma and multiple myeloma (18,19). Based on the literature, however, there are no studies evaluating the relationship between the HALP score and the prognosis of MDS patients. Also , numerous promising biomarkers have been evaluated as potential prognosis predictors for MDS. For instance, low absolute lymphocyte count (ALC) and absolute monocyte count (AMC) levels, decreased serum ApoA1 levels, as well as an increase in the number of mature monocytes in the bone marrow can predict poor prognosis in MDS.(6-9 )However, none of these markers have been adopted into IPSS-R. In recent years, it has also been reported that high FIB is a poor prognostic factor in some tumors.(10-12 )However, evidence of the role of FIB in MDS is lacking. In addition, AST/ALT ratio could be a simple and economic prognostic indicator for MDS and be used as a supplement to IPSS-R, especially when lacking of karyotype or mutation data.

ELIGIBILITY:
Inclusion Criteria:

* • Adults (≥18 years old) diagnosed with MDS according to WHO criteria

  * Availability of complete medical records including laboratory data for hemoglobin, albumin, lymphocyte count, platelet count, monocyte count, fibrinogen level, AST and ALT
  * Patients who were followed for at least 12 months post-diagnosis or until death

Exclusion Criteria:

* Patients with active infections, liver cirrhosis, chronic inflammatory diseases, or concurrent malignancies at time of diagnosis
* Incomplete laboratory or clinical data
* Patients lost to follow-up within less than 3 months of diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years old) diagnosed with MDS according to WHO criteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-01-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
prognostic significance of many factors in MDS | Two years
  to investigate prognostic significance of many factors in MDS including HALP score ( haemoglobin level, albumin level, lymphocyte, platelets), in patients with MDS at Assiut University Hospital HALP : a derived value from a formula: Hemoglobin (g/L) × Albumin (g/L) × Lymphocytes (/L) / Platelets (/L)